CLINICAL TRIAL: NCT01486706
Title: Efficacy and Safety of Gabapentin in Treating Overactive Bladder
Acronym: OAB
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Michael E. Chua (Other)
Collaborators: St. Luke's Medical Center, Philippines (Other)
Responsible Party: Sponsor-Investigator, Michael E. Chua, Medical Doctor, St. Luke's Medical Center, Philippines
Organization: St. Luke's Medical Center, Philippines (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SLMC10-010
Record Dates: First submitted 2011-12-04; First posted 2011-12-06 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Urinary Urgency; Urinary Frequency; Nocturia; Incontinence; Detrusor Uninhibited Activity; Quality of Life
Keywords: Overactive Bladder; Gabapentin; Quality of Life; Urodynamic; safety; Efficacy
MeSH Terms: conditions — Nocturia; Urinary Bladder, Overactive | interventions — Gabapentin; Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Gabapentin (Experimental): Two to three months of behavioral therapy prior to start of Gabapentin 100mg/capsule, initially 1 capsule once a day for 1 week then titrate dosage according to symptoms until maximum dose of 1500mg/day Placebo tablet of Solifenacin Succinate will titrate dose same as Solifenacin arm according to symptoms of patient
  Interventions: Drug: Gabapentin
- Solifenacin Succinate (Active Comparator): Two to three months of behavioral therapy prior to Solifenacin Succinate 5mg/tablet initially 1 tablet once a day then titrate dosage according to symptoms upto maximum dose of 10mg/day Placebo form of Gabapentin will titrate dosage same as Gabapentin group according to symptoms of patient
  Interventions: Drug: Solifenacin Succinate
- Placebo (Placebo Comparator): Two to three months of behavioral therapy prior to Placebo form of Gabapentin and Solifenacin and titrate accordingly same as the treatment arms
  Interventions: Drug: Placebo drugs

INTERVENTIONS:
Drug: Gabapentin — 100mg/capsule initially one capsule once a day then titrate according to the symptoms of the patient upto maximum dose of 1500mg/day
  Arms: Gabapentin
Drug: Solifenacin Succinate — 5mg/tablet initially 1 tablet once a day then titrate up to maximum dose of 10mg/tab
  Arms: Solifenacin Succinate
Drug: Placebo drugs — will titrate medications similar to the active drug group
  Arms: Placebo

SUMMARY:
Overactive bladder (OAB) syndrome as defined by International Continence Society is a pathological condition characterized by irritative symptoms: urinary urgency, with or without incontinence, urinary frequency and nocturia. The syndrome often seriously compromises the quality of life of the patients. The etiology of the OAB is considered multifactorial. Neural plasticity of bladder afferent pathways is one of the proposed mechanisms of OAB. The detrusor muscle itself has for many years been the target for drug treatment such as antimuscarinics. However, depression of detrusor contractility, may results in a reduced ability to empty the bladder and lead to some sympathetic adverse effects, which limits the treatment of OAB. Currently the focus of OAB treatment has changed to other bladder structures/mechanisms, such as afferent nerves and urothelial signaling as targets for intervention. C-fiber bladder afferents nerves may be critical for symptom generation in pathologic states such as OAB because these fibers demonstrate remarkable plasticity. Up-regulation of bladder C-fiber afferent nerve function may also play a role in urge incontinence, overactive bladder (OAB) and sensory urgency. The mechanism of Gabapentin's action for neuropathic pain has not been fully elucidated but is appears to have inhibitory activity on afferent C-fibers nerve activity; moreover, several studies had established the safety of Gabapentin in its treatment of different conditions. Due to the proposed mechanism, the investigators suggest that Gabapentin may be a new alternative for treating OAB.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory and able to use the toilet without difficulty
* History of OAB symptoms for ≥ 3 months
* An average of ≥ 8 micturitions per 24 hours and ≥ 1 urgency episode (with or without incontinence) per 24 hours as documented in a 3-day micturition diary
* Subjects are bothered by symptoms as reflected by OAB-questionnaire

Exclusion Criteria:

* Patient has stress or mixed incontinence
* Patient has Benign Prostatic Hyperplasia with severe lower urinary tract symptoms based on IPSS score
* Patient has uncontrolled Diabetes Mellitus Type II Patient has Diabetes Insipidus, UTI
* Patient has history of interstitial cystitis, painful bladder syndrome, or chronic pelvic pain
* Patient has a history of stroke, seizures, or major neurological disorders
* Patient has a history of fecal incontinence and or continual urine leakage
* Patient has had surgery to correct stress urinary incontinence or pelvic organ prolapse within 6 months of study start
* Patient received bladder training of electrostimulation within 2 weeks of study start
* Patient requires a catheter
* Patient is taking medications that cannot be stopped for the duration of the trial including certain anticholinergics or smooth muscle relaxants
* Patient began taking tricyclic antidepressants, serotonin/norepinephrine reuptake inhibitors, calcium channel blockers, ephedrine/pseudoephedrine, or diuretic therapy less than 8 weeks before study start
* Patient has been on hormone replacement therapy for less than 12 weeks at study start
* Patient must take medication for arrhythmia, contraindicated for Solifenacin or Gabapentin
* Patient has multiple and/or severe allergies to foods and drugs
* Patient regularly uses any illegal drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2010-10; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
improvement of symptom domain means decreased frequency to less than 8 micturitions per 24 hours, no urgency noted per 24 hrs and less that 3 wakening at bedtime for micturation. | 12 weeks
  Mean number of Micturations per 24 hrs, Mean number of urgency episodes pe 24 hrs, mean urgency incontinence episodes per 24hrs and mean nocturia episodes per 24hrs

SECONDARY OUTCOMES:
Improvement of bladder function domain means increased bladder capacity (MVV) | 12 weeks
Improvement in quality of life domain means increased overall quality of life as perceived and result in OAB-q | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marcelino L Morales JR, MD, Study Director — Institute of Urology, St. Luke's Medical Center, Philippines
Locations (1):
- Comprehensive Pelvic Floor Center- St. Luke's Medical Center, Quezon City, National Capital Region, Philippines

REFERENCES:
- [Derived] Chua ME, See MC 4th, Esmena EB, Balingit JC, Morales ML Jr. Efficacy and Safety of Gabapentin in Comparison to Solifenacin Succinate in Adult Overactive Bladder Treatment. Low Urin Tract Symptoms. 2018 May;10(2):135-142. doi: 10.1111/luts.12152. Epub 2017 Feb 2. PMID 28150436